CLINICAL TRIAL: NCT03931148
Title: Feasibility Study of the Interest of Functional Neuroimaging in Assessing Decision-making Capacity of Older People With Neurocognitive Disorders
Brief Title: Interest of Functional Neuroimaging in Assessing Decision-making Capacity of Older People With Neurocognitive Disorders
Acronym: IMAGISION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Principal Investigator, Thomas TANNOU, University Hospital Practitioner, Centre Hospitalier Universitaire de Besancon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: API/2018/100; API3A2018 (Other Grant/Funding Number: CHU de Besancon); Don Du Souffle 2018 (Other Grant/Funding Number: Don du Souffle Besancon); Prix H Mutuelle Alzheimer 2019 (Other Grant/Funding Number: Harmonie Mutuelle - Fondation de l'Avenir)
Record Dates: First submitted 2019-04-23; First posted 2019-04-30 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Decision Making; Dementia; Aging
Keywords: Neuroimaging; Dementia; Decision making; Neuropsychology; Aging
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Masking Description: Analyses of functional imaging results (MRI and/or EEG) will be carried out blindly from the results of the geriatric assessment of decision-making ability. The results between the geriatrician's assessment of decision-making ability and the results of functional imaging tests will then be compared.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): After first consultation for diagnosis of neurodegenerative disorder :
  * Geriatric Assessment with specific neuropsychologic tests of decision making
  * fRMI
  * EEG High Resolution
  * Qualitative interview
  Interventions: Diagnostic Test: Geriatric Assesment with neuropsychological test more specific on decision making; Diagnostic Test: Functional RMI; Diagnostic Test: High Resolution EEG; Other: Qualitative interview

INTERVENTIONS:
Diagnostic Test: Geriatric Assesment with neuropsychological test more specific on decision making — The following tests will be made : MoCA, FAB, TMT, Stroop-Victoria, JAT
Diagnostic Test: Functional RMI — With specific test of decision making (IGT) specially adapted to the population
Diagnostic Test: High Resolution EEG — With specific test of decision making (BART) specially adapted to the population
Other: Qualitative interview — Qualitative semi-directed interviews with participants, their caregivers and their geriatrician to analyse everyday life decision making ability.

SUMMARY:
IMAGISION aims to explore, in a cohort of patients referred for geriatric consultation for neurocognitive evaluation, the contribution of functional neuroimaging (functional MRI and, if possible, high resolution EEG) to geriatric expertise, associated with the performance of a battery of neuropsychological tests in the evaluation of decision-making capacity.

DETAILED DESCRIPTION:
It is during aging of patients, especially those with polypathological disorders and in whom cognitive disorders appear, that the most complex and ethical questions arise. In this context, these patients are frequently referred to geriatric consultations or memory centres for a global assessment of their cognitive functions and life skills in order to optimize their care and anticipate their medical and medico-social future. The assessment of decision-making capacity is essential in this regard.

Nevertheless, there is no test that specifically explores this issue and, therefore, people's decision-making abilities may not be properly estimated and may prevent some patients from making decisions when they would be able to do so.

Thus, although the issue of decision-making has generally been explored from a neuropsychological perspective in many studies, there is no specific test or score for decision-making capacity, as it is a complex process. The question of decision-making capacity in complex situations is therefore addressed by a multiple analysis of many parameters, including different neuropsychological data, which are then synthesized by the clinician in a standardized geriatric assessment to get an idea, among other things, of the overall ability to make decisions.

Given the difficulty of this and the ethical and societal issue, the research question focuses on the contribution of neuroimaging technologies to the assessment of decision-making capacity.

In fact, several studies have explored the issue as part of the functional neuroimaging study. The investigators note, in particular:

* Decision-making studies were conducted using the EEG-High Resolution (EEG-HR) technique. It is a technique for electromagnetic analysis of brain functions with excellent temporal resolution and quite good spatial resolution. This allows, during functional decision tests, a detailed analysis of the temporality of the activation of the frontal and prefrontal areas.
* Functional MRI (fMRI) is a neurological imaging technique whose main strength lies in its spatial acuity. Thus, the performance of functional decisional tests under functional MRI allows a detailed analysis of the recruitment of the different zones between the dorsolateral prefrontal cortex and the median ventromedian cortex.

These 2 neuroimaging techniques allowed a neuro-functional analysis of decision making, based on the realization of more specific tests, modelling decision making. Among these models, the Iowa Game Task and the Balloon Assessement Risk Task are frequently used.

Nevertheless, all these tests and explorations were conducted independently, and no studies have investigated the contribution of a neurofunctional approach to patient decision-making through complementary explorations in functional MRI and /or in EEG-HR as diagnostic tools as part of an overall gerontological evaluation of decision making ability.

The question that arises is therefore that of the development of diagnostic tools.

ELIGIBILITY:
Inclusion Criteria:

* French speaker
* Recent diagnosis of neurocognitive disorder
* Agreed with the study

Exclusion Criteria:

* Delirium
* Major depressive symptoms
* MRI contraindication

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2020-01-05 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Estimation of concordance/disordance between the standardized global gerontological evaluation and the objectification of the activation zones of prefrontal ventromedial and dorsolateral cortex by functional imaging | 1
  The cohort data will be compared between patients identified as " questionable ability " according to the clinical evaluation (reference) and the neuroimaging evaluation, in order to see if the imaging allows to reclassify patients as " able ". A 10 % diagnostic gain in expected.
  Concerning functional neuroimaging (Balloon Analog Risk Task): The lack of activation of specific brain areas during period of interest will be considered as "compatible with the ability to make decisions" on neuro-functional imaging, while patients who do not activate the ROIs in the same situation will be considered as "compatible with questionable decision-making ability".
  Concerning standardized geriatric assessment: At the end of the initial consultation, based on his clinical examination, interview and standardized neuropsychological assessment, the geriatrician will classify each patient either as " preserved decision-making ability " or " questionable decision-making ability ".

OTHER OUTCOMES:
Comparison between neuropsychological test and neurofunctional imaging | 1 day
  The results of the functional neuroimaging tests will be analyzed in comparison with the neuropsychological tests performed, to verify the correlation between the results of the neuropsychological tests of decision-making ability and the results of the neuroimaging tests, and thus to identify, among the battery of tests used, those that are the most discriminating in the evaluation of decision-making ability
Comparison between neurocognitive disorders stage and decision-making ability | 1 day
  The neuropsychological tests that will be carried out will allow to identify the stage of neurocognitive disorders in patients. These elements can be correlated with the analysis of decision-making abilities in order to demonstrate a correlation between neurocognitive disorders, their stage, and decision-making ability
Analysis of the implication of the decision-making ability in everyday life situation | 1 day
  Based on the semi-directed interviews, a qualitative analysis will be carried out to study the reality of everyday life situations where decision-making ability is mobilized. A particular focus will be made on the impact of neurocognitive disorders on aging in place, and thus on the decision to integrate a nursing home.

CONTACTS AND LOCATIONS:
Overall Officials: Regis AUBRY, PhD, Study Chair — Centre Hospitalier Universitaire de Besancon
Locations (2):
- CRIUGM, Montreal, Quebec, Canada
- Centre Hospitalier Universitaire de Besancon, Besançon, Bourgogne-Franche-Comté, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tannou T, Godard-Marceau A, Joubert S, Daneault S, Kergoat MJ, Magnin E, Comte A, Gabriel D, Vidal C, Pazart L, Aubry R. Added value of functional neuroimaging to assess decision-making capacity of older adults with neurocognitive disorders: protocol for a prospective, monocentric, single-arm study (IMAGISION). BMJ Open. 2021 Sep 29;11(9):e053549. doi: 10.1136/bmjopen-2021-053549. PMID 34588264